CLINICAL TRIAL: NCT05290298
Title: Short-term Intervention With Nitrate-based Nutritional Formula on Oxygen Saturation and Patient-reported Outcomes in Covid-19 Patients
Brief Title: Nitrate-based Nutritional Formula for Oxygen Saturation and Patient-reported Outcomes in Covid-19
Acronym: COVID-NITRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Principal Investigator, Sergej Ostojic, Head of Applied Bioenergetics Lab, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-TLI/2021-2
Record Dates: First submitted 2022-03-21; First posted 2022-03-22 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Nitrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NITRATE (Experimental): Multi-component nutritional formula (containing 1200 mg of potassium nitrate, 200 mg of magnesium, 50 mg of zinc, and 1000 mg of citric acid)
  Interventions: Dietary Supplement: NITRATE
- PLACEBO (Placebo Comparator): Placebo (2.5 grams of inulin)
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: NITRATE — Multi-component nutritional formula
  Arms: NITRATE
Dietary Supplement: PLACEBO — Placebo
  Arms: PLACEBO

SUMMARY:
A preliminary open-label case report demonstrated the beneficial effects of an innovative nitrate-based nutritional formula on oxygen saturation in patients with COVID-19. Whether these initial findings are relevant in a more robust research design currently remains unknown. Therefore, the main objective of this randomized controlled trial was to analyze the acute effects of nitrate-based nutritional formula on peripheral SpO2, patient-reported outcomes, and safety indices in patients with acute COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* age 3 18 years
* confirmed SARS-CoV-2 infection
* SpO2 < 95%
* COVID-19 patients in stable condition (i.e., not requiring hospital admission)

Exclusion Criteria:

* regnant or lactating women
* concomitant pulmonary and cardiovascular conditions
* history of dietary supplement use during the past four weeks
* participation in another COVID-19-related study
* unwillingness to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Change in oxygen saturation | Baseline vs. 72 hours post-intervention
  Measured at baseline and 72 hours post-intervention

SECONDARY OUTCOMES:
Change in fatigue | Baseline vs. 72 hours post-intervention
  Measured at baseline and 72 hours post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostojic SM, Milovancev A, Drid P, Nikolaidis A. Oxygen saturation improved with nitrate-based nutritional formula in patients with COVID-19. J Int Med Res. 2021 Apr;49(4):3000605211012380. doi: 10.1177/03000605211012380. PMID 33906526